CLINICAL TRIAL: NCT06636994
Title: Anatomical and Functional Predictions of Blindsight Capabilities in Post-Stroke Patients With Homonymous Hemianopia (PRE-SIGHT)
Brief Title: Anatomical and Functional Predictions of Blindsight Capabilities in Patients With Lateral Hemianopsia
Acronym: PRE-SIGHT
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CGC_2024_3
Record Dates: First submitted 2024-08-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Homonymous Hemianopia; Stroke; Cortical Blindness; Hemianopia
MeSH Terms: conditions — Hemianopsia; Stroke; Blindness, Cortical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Homonymous lateral hemianopia (HLH) is characterized by loss of vision in half the visual field, and is the most common neurovisual disorder following stroke.

Numerous behavioral and neuroanatomical studies have focused on the phenomenon of blindsight, corresponding to patients' unconscious residual visual capacities in the blind hemifield. Cohort studies of patients have highlighted different types of blindsight, and a low occurrence of the phenomenon initially described: (1) type 1 blindsight (≈12%), unconscious visual abilities; (2) type 2 blindsight, visual abilities associated with sensations in the blind field (≈18%); (3) blindsense, sensations in the blind field without visual abilities (≈30%); and (4) no blindsight (≈40%). The heterogeneity of these blindsight abilities in the HLH population is closely related to patients' neuroanatomical and functional profiles.

In particular, resting-state functional imaging (r-fMRI) and default mode network analysis have highlighted a significant correlation between the degree of inter-hemispheric connection (between the healthy and injured hemispheres) and the rate of spontaneous visual field recovery. To our knowledge, this degree of functional connectivity has not yet been studied in relation to blindsight abilities. However, this functional MRI measurement tool represents a potential predictive factor for patients' residual performance in their blindsight field, in order to assess the level of visuo-cognitive impairment and, ultimately, to adapt care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and over
* with homonymous visual field amputation sequelae of a retrochiasmatic lesion of vascular origin (stroke), including the occipital region (primary visual cortex, optic radiations, associated occipital areas)
* Requires follow-up brain MRI as part of treatment
* Able to perform experimental tasks on computer
* Express consent to participate in the study
* Member or beneficiary of a social security scheme

Exclusion Criteria:

* Severe neuropsychological disorders (language, memory, attention, vigilance, reasoning)
* Severe ophthalmological disorders or visual acuity below 3/10 prior to stroke
* Progressive ophthalmological disorders (cataract or glaucoma) likely to bias measurements
* Major psychiatric or behavioral disorders making care impossible
* Patient benefiting from a legal protection measure
* Pregnant or breast-feeding women (declarative information)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with homonymous lateral hemianopia undergoing cerebral MRI for follow-up and rehabilitation following stroke
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Description of resting-state functional MRI measurement of the degree of Resting State Functional Connectivity (RSFC) between left and right hemisphere regions. | DAY 0
  Comparison of the degree of inter-hemispheric Resting State Functional Connectivity between the four patient groups: absence of blindsight, type I blindsight, type II blindsight and blindsense.

SECONDARY OUTCOMES:
Correlation between inter-hemispheric functional connectivity and blindsight performance | DAY 0
  Resting-state functional MRI measurement of the degree of RSFC between left and right hemisphere regions of interest.
  Blindsight performance assessed by measuring the sensitivity of discrimination of spatial orientation (horizontal/vertical) of lines presented in the patient's blind field (blindsight).
Density and intensity of visual and attentional default networks in each type of blindsight | DAY 0
  Calculation (Graph Theory) of neural network matrices, weighted and created on the basis of correlations of activations in different brain regions during resting-state functional MRI measurement .
Blindsight performance according to the laterality of the lesion (left or right hemisphere) | DAY 0
  Blindsight performance assessed by measuring the sensitivity of discrimination of spatial orientation (horizontal/vertical) of lines presented in the patient's blind field (blindsight)
Correlation between the level of inter-hemispheric functional connectivity and blindsight performance | DAY 0
  Resting-state functional MRI measurement of the degree of Resting State Functional Connectivity (RSFC) between left and right hemisphere regions of interest, blindsight performance assessed by measuring the sensitivity of spatial orientation discrimination (horizontal/vertical) of lines presented in the blindsight field.
Correlation between visual default network density and intensity and blindsight performance | DAY 0
  Computation (Graph Theory) of neural network matrices, weighted and created on the basis of correlations of activations of different brain regions during Resting-state functional MRI measurement. Blindsight performance assessed by measuring the sensitivity of discrimination of spatial orientation (horizontal/vertical) of lines presented in the patient's blind field (blindsight).
Correlation between lesion volume and blindsight performance | DAY 0
  Blindsight performance assessed by measuring the sensitivity of spatial orientation discrimination (horizontal/vertical) of lines presented in the patient's blind field (blindsight).

CONTACTS AND LOCATIONS:
Overall Officials: Clémentine GARRIC, Principal Investigator — Integrative Neuroscience and Cognition Center
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France